CLINICAL TRIAL: NCT02658474
Title: Multidisciplinary Group Based Treatment of Patients With Chronic Pain. A Randomized Controlled Trial Comparing Acceptance Commitment Therapy and Treatment in a Primary Care Setting
Brief Title: Multidisciplinary Group Based Treatment of Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1880REK
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Acceptance and Commitment Therapy; Multidisciplinary treatment; Group treatment
MeSH Terms: conditions — Chronic Pain | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT-group (Experimental): Group based Acceptance and Commitment Therapy. The patients will attend to three sessions which last for three days. Between the sessions the patients will train at home on ACT related topics. The whole intervention will last for three months.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Primary care (No Intervention): Treatment in a primary care setting.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Group based Acceptance and Commitment Therapy
  Arms: ACT-group

SUMMARY:
The purpose of this study is to determine whether group based Acceptance and Commitment Therapy (ACT) at a university hospital clinic is superior to treatment in a primary care setting among patients with chronic pain.

Hypothesis:

i) A group based ACT treatment leads to less pain and greater Health Related Quality of Life (HRQOL) in patients with chronic pain than treatment in a primary care setting.

ii) The improvement in pain and HRQOL is mediated through an increased degree of pain willingness and involvement in activities.

iii) Improvement of pain and HRQOL after the two treatments is associated with demographic, psychosocial and somatic characteristics.

DETAILED DESCRIPTION:
Background:

Chronic pain represents a substantial social problem. In Norway, the prevalence of chronic moderate pain is between 25 and 30%, and for severe pain it is at 2%. Multidisciplinary treatment is recommended for chronic pain, and during the last years Acceptance Commitment Therapy (ACT) has been implemented.

Research design, methods and analyses:

One hundred and twenty participants will be recruited from a list of patients referred to the Multidisciplinary Pain Department at the University Hospital of North Norway. Those who meet the defined criteria, are invited to participate. The study has a randomized, semi-crossover design. The participants are allocated to group based ACT or treatment in a primary care setting with a gender stratified, block randomization with a ratio of 1: 1. This means that half of the participants (intervention group, n: 60) get early group based ACT, while the other half (control group, n: 60) will be treated in a primary health care setting. Those of the control group who still meet the criteria, will be offered ACT afterwards.

Data collection will take place at a) start of the study, b) a few days prior to the onset of ACT and c) a few days after ended ACT, and 6 months after the onset of ACT. Data collection is carried out with the same time intervals in the control group. After having received ACT data is collected 12 months after the onset of ACT.

Treatment protocol:

At the first appointment all participants undergo a multidisciplinary evaluation where participants alternate between telling their life story and listening to responses from the multidisciplinary team. The aim is to initiate a reflexive attitude and a feeling of being acknowledged. The multidisciplinary report to the general practitioner provides diagnostic considerations as well as recommendations for future treatment.

A. Intervention group: Acceptance Commitment Therapy (ACT) is based on the principles of operant conditioning and is less problem-oriented compared with Cognitive Behavioral Therapy (CBT). The patients learn how to accept and to realize that thoughts, feelings and sensations do not have to decide how life is. In a comparative efficacy study ACT has been shown equally effective as CBT.

Mindfulness Based Stress Reduction is included in ACT, and the patients will therefore get a systematic training in mastering stress and emotional conflicts.

B: Control Group: Patients in the control group are primarily treated by the general practitioner supported by recommendations from the multidisciplinary pain team. The treatment will vary in content and form.

Variables:

Electronic data storage: Data will be collected by an internet based system according the the Norwegian regulations for social insurance and are imported and stored anonymized in a password protected SPSS file data at the University Hospital of North Norway.

Variables:

The demographic variables include gender, year of birth, marital status, number of children, education, occupation and employment status, as well as benefits from the social security system (NAV), financial situation and possible compensation or application for disability.

Clinical variables include comorbidity specified by a list of diseases related to the major organ systems.

Pain analyses: Pain intensity is one of two primary outcomes and is measured with four numerical scales for pain intensity (0 being no pain and 10 the worst possible pain) obtained from the Brief Pain Inventory. Localization (specified by a body map) and temporal aspects, duration and variety of pain are also measured

Health related Quality of life: Short form 36 (version 2).

Physical activity: The Gothenburg Activity Question .

Sleep: Insomnia Severity Index is a self-reporting questionnaire that assesses the severity of the sleeping problems. The form contains seven questions answered with a 5 point Likert scale.

Fatigue: Chalder fatigue questionnaire contains 11 questions and operates with 4 answer options with varying degrees of severity.

Anxiety and depression: Hopkins Symptom Checklist 25 with 25 questions about anxiety and depression.

Pain catastrophizing: The Pain Catastrophizing Scale with 13 questions measuring rumination, worst case thinking and helplessness. General Self-Efficacy: General Perceived Self-Efficacy Questionnaire is based on Bandura's model.

Adverse life events: Those who report positively on a severe life event are asked to fill in Impact of Event Scale-6 with 6 questions related to thoughts after traumatic life event.

Specific evaluation of the ACT intervention: The questionnaire Chronic Pain Acceptance Questionnaire (CPAQ 20) includes 20 items selected to assess the degree of pain willingness and involvement in relation to activities.

Use of health services: Type and number of treatments given in and outside the Pain department with waiting time and expectations to treatment.

Drug Consumption: Consumption of non-opioids (paracetamol and NSAIDs), opioids (daily dose is converted to morphine equivalents), and coanalgesics (antidepressants and anticonvulsants) are recorded by a physician.

Statistics: The investigators will perform repeated comparisons of the two treatment groups over a 6 month period, and "within-group" comparisons of ACT treated patients over a 12 month period. The statistical analyses will be carried out in collaboration with a statistician. Comparison analyses between the groups and to baseline as well as predictor analyses will be performed by Mixed models (SPSS).

Power: Based on previously published studies and power calculations from pilot data, a statistical power of 80% and significance level of 5% the investigators will include 120 patients.

Project plan, project, organization and Cooperation:

The project is an independent part in a national multicenter survey of patients treated at multidisciplinary pain departments at university hospitals in Norway. Our project will largely use the same screening measures and outcomes as the national survey.

Ethics: This study compares two established therapy modalities offered to patients referred to the Pain department at the University Hospital of North Norway. The project was approved by the Regional Committee for Medical and Health research ethics 10/12/13.

ELIGIBILITY:
Inclusion Criteria:

* Long-term pain condition over 6 months.
* Strongest pain ≥ 4 on a scale of 0 to 10.
* Consent competent and over 18 years
* Motivated for group-based psychological (ACT) treatment.

Exclusion Criteria:

* Psychiatric illness and behavioral problems, including substance abuse that prevents good group interaction
* Severe progressive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-08; Primary Completion 2021-10-02 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Group difference in pain intensity | 3 months after baseline
  Continuous variable (Numeric rating scale) analyzed by Mixed Model
Group difference in pain intensity | 6 months after baseline
  Continuous variable (Numeric rating scale) analyzed by Mixed Model
Group difference in health related quality of life | 3 months after baseline
  Health related quality of life is measured by Short Form-36 and analyzed by Mixed Model
Group difference in health related quality of life | 6 months after baseline
  Health related quality of life is measured by Short Form-36 and analyzed by Mixed Model

SECONDARY OUTCOMES:
Change from baseline in pain intensity | 3 months after baseline
  Continuous variable (Numeric rating scale) analyzed by Mixed Model
Change from baseline in pain intensity | 6 months after baseline
  Continuous variable (Numeric rating scale) analyzed by Mixed Model
Change from baseline in pain intensity | 12 months after baseline
  Continuous variable (Numeric rating scale) analyzed by Mixed Model
Change from baseline in health related quality of life | 3 months after baseline
  Health related quality of life is measured by Short Form-36 and analyzed by Mixed Model
Change from baseline in health related quality of life | 6 months after baseline
  Health related quality of life is measured by Short Form-36 and analyzed by Mixed Model
Change from baseline in health related quality of life | 12 months after baseline
  Health related quality of life is measured by Short Form-36 and analyzed by Mixed Model
Change from baseline in pain willingness and involvement in activities | 3 months after baseline
  The questionnaire Chronic Pain Acceptance Questionnaire (CPAQ 20) and analyzed by Mixed Model
Change from baseline in pain willingness and involvement in activities | 6 months after baseline
  The questionnaire Chronic Pain Acceptance Questionnaire (CPAQ 20) and analyzed by Mixed Model
Change from baseline in pain willingness and involvement in activities | 12 months after baseline
  The questionnaire Chronic Pain Acceptance Questionnaire (CPAQ 20) and analyzed by Mixed Model
Group difference in drug consumption | 6 months after baseline
  Number of analgesics and morphine equivalents analyzed by Mixed Model
Group difference in consumption of health services | 6 months after baseline
  Number of health services applied is counted and analyzed by Mixed Model

CONTACTS AND LOCATIONS:
Overall Officials: Gunnvald Kvarstein, PhD, Principal Investigator — UiT The Arctic University of Tromsø
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No